CLINICAL TRIAL: NCT00325117
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study to Compare the Effect of 12 Weeks Treatment With Vildagliptin to Placebo as Add-on Therapy to Sulfonylurea in Patients With Type 2 Diabetes Inadequately Controlled With Sulfonylurea Monotherapy
Brief Title: To Assess the Efficacy and Safety of Vildagliptin as Add-on Therapy to Sulfonylurea in Patients With Type 2 Diabetes Inadequately Controlled With Sulfonylurea Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A1302
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2007-05-14 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Vildagliptin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is not being conducted in the United States. Vildagliptin is an oral antidiabetic agent. This 12-week clinical study is designed as a multicenter, randomized, double-blind, parallel-group, placebo-controlled study aimed to evaluate the efficacy and safety of vildagliptin as add-on therapy to a sulfonylurea in patients with type 2 diabetes inadequately controlled with sulfonylurea monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes and treated with a stable dose of sulfonylurea
* Patients on diet and exercise who have not reached target blood glucose levels
* Outpatients

Exclusion Criteria:

* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant cardiovascular complications as defined by the protocol
* Significant diabetic complications as defined by the protocol

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-04

PRIMARY OUTCOMES:
Change from baseline to endpoint on HbA1c at 12 weeks

SECONDARY OUTCOMES:
Change from baseline to endpoint on fasting plasma glucose at 12 weeks
Change from baseline to endpoint in HOMA B at 12 weeks
Change from baseline to endpoint in HOMA IR at 12 weeks
Change from baseline to endpoint on fasting lipids at 12 weeks
Adverse events profile after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan

REFERENCES:
- [Derived] Kikuchi M, Haneda M, Koya D, Tobe K, Onishi Y, Couturier A, Mimori N, Inaba Y, Goodman M. Efficacy and tolerability of vildagliptin as an add-on to glimepiride in Japanese patients with Type 2 diabetes mellitus. Diabetes Res Clin Pract. 2010 Sep;89(3):216-23. doi: 10.1016/j.diabres.2010.04.017. PMID 20537746